CLINICAL TRIAL: NCT01876121
Title: Celecoxib Japan Observational Study for the Patients With Acute Pain
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: COX-05
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Patients With Traumatic Pain, Post-surgical Pain and Tooth Extract Pain
Keywords: NSAIDs; Acute pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Celecoxib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Celecox group
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib — oral
  Other Names: Celecox

SUMMARY:
This study is to assess the safety and efficacy of celecoxib on the pain relief from acute pain.

DETAILED DESCRIPTION:
Patients with traumatic pain, post-surgical and tooth extract pain will be included in this study. Patients will receive Celecoxib for 2 weeks and the efficacy on pain relief and the safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with traumatic pain, post-surgical pain and tooth extract pain

Exclusion Criteria:

* Hyperreactive to sulfonamide
* Aspirin asthma patients
* Peptidic ulcer patients
* Serious liver disease patients
* Serious kidney disease patients
* Serious heart failure patients
* End of pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with traumatic pain, post-surgical pain and tooth extract pain
Sampling Method: Non-Probability Sample
Enrollment: 784 (Actual)
Dates: Start 2012-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety assessed by the incidence of adverse events and lab-tests | For 2 weeks

SECONDARY OUTCOMES:
Overall pain improvement assessed by visual analogue scale (VAS) | Baseline and week-2

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Shikoku
  - Tōhoku